CLINICAL TRIAL: NCT00283712
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Infliximab in Subjects With Pemphigus Vulgaris Receiving Prednisone
Brief Title: Use of Infliximab for the Treatment of Pemphigus Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT APV01
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Pemphigus
Keywords: Skin Diseases; Autoimmune Diseases
MeSH Terms: conditions — Pemphigus; Skin Diseases; Autoimmune Diseases | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Infliximab (Experimental): Participants are randomized to receive intravenous infusions of infliximab (5mg/kg reconstituted in 10 mL of Sterile Water for Injection, USP ) at Weeks 0, 2, 6, and 14 over a time period of no less than two hours in a masked (blinded) fashion. Refer to section titled, "Detailed Description" for additional treatment information.
  Interventions: Drug: Infliximab
- Placebo Comparator (Placebo Comparator): Participants are randomized to receive intravenous infusions of placebo (5 mg/kg comprised of a white lyophilized powder reconstituted in 10 mL of Sterile Water for Injection, USP) at Weeks 0, 2, 6, and 14 over a time period of no less than two hours in a masked (blinded) fashion. Refer to section titled, "Detailed Description" for additional treatment information.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Infliximab — Chimeric IgG monoclonal antibody that binds to TNF-alpha, generally used to treat Crohn's disease, given in a dosage of 5 mg/kg
  Other Names: Remicade®
  Arms: Infliximab
Other: Placebo Comparator — Placebo administered in place of infliximab for control group
  Other Names: Control Arm
  Arms: Placebo Comparator

SUMMARY:
Pemphigus vulgaris (PV) is a rare skin disorder that causes blistering of the skin and mucous membranes. Infliximab is a man-made antibody used to treat certain types of immune system disorders, including rheumatoid arthritis and Crohn's disease. This study will determine if infliximab given in combination with prednisone is a safe and effective treatment for adults with PV.

DETAILED DESCRIPTION:
PV involves blistering of the outer layer of skin and mucous membranes, causing a separation of epidermal cells. The disease occurs when the immune system produces antibodies to specific proteins in the skin and mucous membranes; the cause for production of these autoantibodies is unknown. Infliximab is a genetically engineered monoclonal antibody directed against tumor necrosis factor (TNF)-alpha, a chemical messenger that activates an immune response. Infliximab has been used to treat other autoimmune disorders, including rheumatoid arthritis, ankylosing spondylitis, and Crohn's disease. This study will evaluate the safety and efficacy of infliximab given in combination with prednisone for the treatment of adults with PV.

This study will last 26 weeks. At study entry, all patients will be taking a stable dose of prednisone (or an equivalent corticosteroid) of 20 to 120 mg/day for at least 2 weeks prior to study entry. Patients will be randomly assigned to one of two arms: experimental or placebo comparator. The experimental treatment arm will receive infusions of infliximab, and the control arm will receive placebo. Infusions will be given at study entry and Weeks 2, 6, and 14. Before the start of each infusion, a physical exam, vital signs measurement, medical and medication history, review of a disease activity log, a skin evaluation, and blood collection will occur. During each infusion and for 1 hour postinfusion, patients' vital signs will be monitored for any adverse events. Patients will need a responsible adult to take them home after they are discharged from the treatment facility; this person should remain with the patient overnight in case any problems arise from the treatment. The patient will be contacted by phone that night and the next morning after infusion and will be asked about any adverse effects they may have experienced. Those patients that experience adverse effects may be asked to return to the treatment facility for examination. Prednisone doses may be tapered by 15 percent every 2 weeks during the study at the investigator's discretion.

There will be a total of 9 study visits until Week 26: screening, study entry, Week 2, and every 4 weeks thereafter. Each study visit will include a physical exam, vital signs measurement, medical and medication history, a review of the disease activity log and adverse events experienced since the last visit, skin assessments, and blood collection; patients will also be asked to complete a tuberculosis (TB) questionnaire. Patients will be asked to complete quality of life questionnaires at study entry and Weeks 10, 18, and 26. Skin biopsies of unaffected skin will be done at study entry and Weeks 10, 18, and 26; if patients have PV-associated lesions, additional skin biopsies of affected skin will be done at study entry and Week 18.

ELIGIBILITY:
Inclusion Criteria:

* Positive direct immunofluorescence of patient's skin showing IgG or complement C3 protein on cell surface with histopathology of lesional skin biopsies consistent with diagnosis of pemphigus vulgaris
* Failure to completely respond to standard steroid therapy (equivalent to prednisone 1 to 2 mg/kg/day followed by tapering)
* Systemic corticosteroid therapy of at least 20 mg prednisone daily and no more than 120 mg/day
* Inability to reduce systemic corticosteroid dosage below 20 mg/day for at least 8 weeks
* Stable dosage of prednisone for at least 2 weeks prior to study entry
* Oral/mucosal disease or skin disease. Detailed information about this criterion can be found in the protocol
* Willing to comply with the study protocol
* Willing to use acceptable means of contraception for the duration of the study and for 6 months after the end of the study

Exclusion Criteria:

* Positive tuberculosis (TB) test within 1 month prior to first administration of study drug
* History of latent or active TB prior to screening
* Signs or symptoms suggestive of TB disease by medical history or physical examination within 3 months prior to first administration of study drug
* Posterior/anterior/lateral chest radiograph within 3 months prior to screening showing evidence of cancer, infection, or abnormalities (apical scarring) suggestive of previous TB
* Serious infection, hospitalization for an infection, or treatment with intravenous (IV) antibiotics for an infection within 2 months prior to screening. Patients who have had less serious infections are eligible for this study at the discretion of the investigator.
* History or presence of opportunistic infections within 6 months prior to screening
* History of receiving human/murine recombinant products
* Known allergy to murine products or other chimeric proteins
* Human immunodeficiency virus (HIV) infected
* Chronic hepatitis B or hepatitis C virus infection
* History of hepatitis C virus infection
* Cancer within the 5 years prior to study entry. Patients with completely resected non-melanoma skin cancers are not excluded.
* History or presence of congestive heart failure
* History or presence of seizure or demyelinating disorder
* History of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis
* Received a Bacillus Calmette-Guerin (BCG) vaccine within 12 months of screening
* History of lymphoproliferative disease, including lymphoma or signs and symptoms of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location or enlarged spleen
* Current signs or symptoms of severe progressive or uncontrolled kidney, liver, blood, gastrointestinal, endocrine, lung, heart, neurologic, or cerebral disease
* Have had chronic or recurrent infectious disease including, but not limited to, chronic kidney infection, chronic chest infection, sinusitis, recurrent urinary tract infection, infected skin wound, or ulcer
* Previous treatment with infliximab, other monoclonal antibodies, or antibody fragments
* Previous treatment with etanercept or other anti-tumor necrosis factor (TNF) agents in the 3 months prior to screening
* Treatment with methotrexate, azathioprine, mycophenolate mofetil, plasmapheresis, IV immunoglobulin, pulse systemic corticosteroids, or other systemic immunosuppressive agents within the 4 weeks prior to study entry
* History of alcohol or drug abuse within the 3 years prior to study entry
* History of noncompliance to medical regimens
* History of a systemic inflammatory disease other than pemphigus vulgaris
* History of a medical condition that would interfere with participation or increase the risk to the participant
* Unable or unwilling to undergo blood draws because of poor tolerability or lack of easy access
* Use of any investigational drug within 30 days prior to screening OR within 5 half-lives of the investigational agent, whichever is longer
* Participation in another investigative clinical trial
* Presence of transplanted solid organ. Participants who have received a corneal transplant more than 3 months prior to screening are not excluded.
* Require certain medications
* Other conditions or circumstances that could interfere with participant's adherence to the study requirements
* Pregnancy, breastfeeding, or plans to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell P. Hall, MD, Study Chair — Division of Dermatology, Duke University Medical Center; E. William St. Clair, MD, Study Chair — Division of Rheumatology and Immunology, Duke University Medical Center; Garnett Kelsoe, DSci, Principal Investigator — Department of Immunology, Duke University; Victoria Werth, MD, Principal Investigator — Department of Dermatology, University of Pennsylvania School of Medicine; Janet Fairley, MD, Principal Investigator — Department of Dermatology, University of Iowa; David Woodley, MD, Principal Investigator — Department of Dermatology, Norris Cancer Center, University of Southern California
Locations (4):
- United States (4):
  - Norris Cancer Center, University of Southern California, Los Angeles, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Anhalt GJ, Diaz LA. Pemphigus vulgaris--a model for cutaneous autoimmunity. J Am Acad Dermatol. 2004 Jul;51(1 Suppl):S20-1. doi: 10.1016/j.jaad.2004.01.011. No abstract available. PMID 15243495
- [Background] Drosou A, Kirsner RS, Welsh E, Sullivan TP, Kerdel FA. Use of infliximab, an anti-tumor necrosis alpha antibody, for inflammatory dermatoses. J Cutan Med Surg. 2003 Sep-Oct;7(5):382-6. doi: 10.1007/s10227-002-0134-1. Epub 2003 Sep 24. PMID 14973643
- [Background] Jacobi A, Shuler G, Hertl M. Rapid control of therapy-refractory pemphigus vulgaris by treatment with the tumour necrosis factor-alpha inhibitor infliximab. Br J Dermatol. 2005 Aug;153(2):448-9. doi: 10.1111/j.1365-2133.2005.06744.x. No abstract available. PMID 16086769
- [Background] Pardo J, Mercader P, Mahiques L, Sanchez-Carazo JL, Oliver V, Fortea JM. Infliximab in the management of severe pemphigus vulgaris. Br J Dermatol. 2005 Jul;153(1):222-3. doi: 10.1111/j.1365-2133.2005.06672.x. No abstract available. PMID 16029365
- [Result] Hall RP 3rd, Fairley J, Woodley D, Werth VP, Hannah D, Streilein RD, McKillip J, Okawa J, Rose M, Keyes-Elstein LL, Pinckney A, Overington A, Wedgwood J, Ding L, Welch B. A multicentre randomized trial of the treatment of patients with pemphigus vulgaris with infliximab and prednisone compared with prednisone alone. Br J Dermatol. 2015 Mar;172(3):760-8. doi: 10.1111/bjd.13350. Epub 2015 Feb 5. PMID 25123295
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY655 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY655 — Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. Data analysis tools are also available to researchers.
- Available data/document: Study Protocol: SDY655 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY655 — ImmPort study identifier is SDY655
- Available data/document: Study summary, -design, -adverse event(s), -summary of participant assessments, -interventions, -medications, -demographics, -lab tests, -mechanistic Assays, -study files et al.: SDY655 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY655 — ImmPort study identifier is SDY655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four study centers in the United States enrolled 20 subjects with pemphigus vulgaris (PV) who met entry criteria between August 2005 and December 2010.
Pre-assignment Details: Each participant signed an informed consent before undergoing any screening procedures to assess eligibility. Refer to the Eligibility Section for further details.
Groups:
- Experimental: Infliximab (Remicade, Revellex): Participants were randomized to receive intravenous infusions of infliximab (5mg/kg reconstituted in 10 mL of Sterile Water for Injection, USP ) at Weeks 0, 2, 6, and 14 over a time period of no less than two hours in a blinded (masked) fashion. Refer to section titled, "Detailed Description" for additional treatment information.
- Placebo Comparator: Placebo: Participants were randomized to receive intravenous infusions of placebo (5 mg/kg comprised of a white lyophilized powder reconstituted in 10 mL of Sterile Water for Injection, USP) at Weeks 0, 2, 6, and 14 over a time period of no less than two hours in a blinded (masked) fashion. Refer to section titled, "Detailed Description" for additional treatment information.
Period: Overall Study
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Started | 10 | 10
Intent-to-treat Sample | 10 | 10
Safety Sample | 10 | 10
Per-Protocol Sample | 6 | 7
Completed | 10 | 9 (One subject in placebo arm died prior to study completion.)
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (15.2) | 51.1 (13.9) | 49.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
PDAI Index Total Score [Mean (Standard Deviation); unit: Total Activity Score] — The Pemphigus Disease Area Index (PDAI) was developed by the International Pemphigus Committee and measures both activity of and damage due to pemphigus on the skin, scalp, and mucous membranes. Total scores can range from 0 to a possible 263 maximum score, with 250 points representing disease activity (120 points for skin activity, 10 points for scalp activity, and 120 points for mucosal activity) and 13 points representing disease damage. Higher scores reflect worse disease.
  Total Activity Score | 23.0 (14.6) | 20.8 (10.7) | 21.9 (12.4)
Pemphigus Vulgaris Disease Activity Score: Mucosal [Number; unit: Participants] — The Pemphigus Vulgaris Disease Activity(PVDA)score was used to grade a participant's baseline disease activity using the SAGE II computerized burn mapping system, which calculated the total body surface area(BSA)involved. Scores were based on the number of lesions and blisters present as well as total body surface area involved. Three types of disease activity were assessed: mucosal, cutaneous, and other organ system. A higher score indicates more severe disease activity. For each of the 3 types of disease activity, the number of participants who met the disease activity condition is shown.
  Participants
    No oral ulcers | 1 | 2 | 3
    1 to 5 lesions, small ulcers | 6 | 2 | 8
    6 to 10 lesions, small ulcers | 2 | 5 | 7
    >10 lesions or extension erosions | 1 | 1 | 2
Pemphigus Vulgaris Disease Activity Score: Cutaneous [Number; unit: Participants] — The Pemphigus Vulgaris Disease Activity(PVDA)score was used to grade a participant's baseline disease activity using the SAGE II computerized burn mapping system, which calculated the total body surface area(BSA)involved. Scores were based on the number of lesions and blisters present as well as total body surface area involved. Three types of disease activity were assessed: mucosal, cutaneous, and other organ system. A higher score indicates more severe disease activity. For each of the 3 types of disease activity, the number of participants who met the disease activity condition is shown.
  Participants
    No blisters or erosions | 3 | 3 | 6
    <20 blisters or <1 to 3% BSA | 2 | 4 | 6
    20 to 40 blisters or 3 to 10% BSA | 4 | 2 | 6
    >40 blisters or >10% BSA | 1 | 1 | 2
Pemphigus Vulgaris Disease Activity Score: Other Organ System [Number; unit: Participants] — The Pemphigus Vulgaris Disease Activity(PVDA)score was used to grade a participant's baseline disease activity using the SAGE II computerized burn mapping system, which calculated the total body surface area(BSA)involved. Scores were based on the number of lesions and blisters present as well as total body surface area involved. Three types of disease activity were assessed: mucosal, cutaneous, and other organ system. A higher score indicates more severe disease activity. For each of the 3 types of disease activity, the number of participants who met the disease activity condition is shown.
  Participants
    No eye, esophageal, laryngeal involvement | 9 | 10 | 19
    Any eye, esophageal, laryngeal involvement | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participant Response to Treatment at Week 18
Description: Participants classified as responders at Week 18 had: 1. Achieved a prednisone dosage <= 25% of the initial starting dose or <= 10 mg/day (whichever is greater), and 2. Had no new blisters within the previous 4 weeks.
Time Frame: Baseline to Week 18
Population: Intent-to-Treat
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1
Statistical Analysis 1: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; The study goals were to gather evidence of safety and possible efficacy of infliximab for treatment of pemphigus vulgaris (PV). The analyses focused on estimation rather than hypothesis testing; therefore, there was not sufficient power to detect plausible treatment differences unless they were very large. The sample size reflects a balance between the desire to meet study goals and to expose as few participants as possible until the safety of infliximab for treatment of PV has been clarified; Test type: Superiority or Other; p = 1.00, Fisher Exact; Risk Difference (RD) = 0.00, 90% CI 2-sided [-0.22 to 0.22]
Statistical Analysis 2: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.00, 90% CI 2-sided [0.02 to 42.67]

2. Primary Outcome: Treatment-Related Adverse Events >= Grade 3 On or Before Week 18
Description: Grades were based on the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0. An adverse event (AE) was considered treatment-related if it was classified as unlikely, possibly, probably, or definitely related to study treatment. Participants who experienced at least one treatment-related, grade 3 or higher AE were counted only once. AEs of skin including rash, skin ulceration, and chelitis as defined by the NCI-CTCAE V3.0 System Organ Class of "Skin and Subcutaneous Tissues Disorders" were excluded.
Time Frame: Baseline to Week 18
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants | 0 | 10
Statistical Analysis 1: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; Test type: Superiority or Other; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.26 to 0.06]

3. Secondary Outcome: Participant Response to Treatment at Week 18
Description: Participants classified as responders at Week 18 had: 1. Achieved a prednisone dosage <= 25% of the initial starting dose or <=10 mg/day (whichever is greater), and 2. Had no new blisters within the previous 4 weeks.
Time Frame: Baseline to Week 18
Population: Per-protocol
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 6 | 7
Participants | 1 | 1
Statistical Analysis 1: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; The primary endpoint analysis was replicated using the per-protocol population; Test type: Superiority or Other; p = 1.00, Fisher Exact — All secondary analyses are considered supplemental supportive analyses; Risk Difference (RD) = 0.02, 90% CI 2-sided [-0.31 to 0.36]
Statistical Analysis 2: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; The primary endpoint analysis was replicated using the per-protocol population; Test type: Superiority or Other; p = 1.00, Fisher Exact — All secondary analyses are considered supplemental supportive analyses; Odds Ratio (OR) = 0.83, 90% CI 2-sided [0.02 to 38.35]

4. Secondary Outcome: Participant Modified Response Status at Week 18
Description: Modified responder status was defined as participants achieving a prednisone dosage <=25% of the initial starting dose or <=10 mg/day (whichever is greater) at Week 18 regardless of status on new blister formation during the previous 4 weeks.
Time Frame: Baseline to Week 18
Population: Intent-to-Treat
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants | 5 | 3
Statistical Analysis 1: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.65, Fisher Exact; Risk Difference (RD) = 0.20, 90% CI 2-sided [-0.15 to 0.55]
Statistical Analysis 2: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.650, Fisher Exact; Odds Ratio (OR) = 0.43, 90% CI 2-sided [0.06 to 2.79]

5. Secondary Outcome: Participant Time to Cessation of New Blisters
Description: Time to cessation of new blisters was defined as the time from a participant's first treatment infusion date to the first date where that date and all subsequent dates had no new blisters. Participant diaries were used to assess new blister formation. To achieve cessation, participants had to be free of new blisters at least 3 weeks prior to their last assessment. In order to analyze missing or incomplete data, the data was censored at the date where a participant had no more data or on the date where 50% of the participant's data was missing past that point.
Time Frame: Baseline to Week 26
Population: Subset of Intent-to-Treat Who Experienced Cessation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 5 | 3
Days | 133.0 (31.7) | 98.0 (49.5)

6. Secondary Outcome: Time to 80% Lesion Healing
Description: Time to 80% healing of existing erosions/ulcerations at time of enrollment was assessed using the SAGE II computerized burn-mapping system. The date of 80% healing of existing erosions/ulcerations at time of enrollment was defined as follows: the first date at which the percent of total body surface area (BSA) involved is at least 80% less than the percent of total BSA calculated at the time of enrollment, where the baseline percent of total BSA must be greater than zero percent. If a participant had missing post-baseline assessments, their data was censored at their last non-missing assessment date.
Time Frame: Baseline to Week 26
Population: Subset of Intent-to-Treat Who Experienced Lesion Healing
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 5 | 4
Days | 77.8 (74.4) | 58.0 (36.0)

7. Secondary Outcome: Total Prednisone Dosage Required for Participants to Achieve Cessation of New Blisters
Description: Each participant's prednisone dose was summed from the time of enrollment until the date of cessation of new blisters. Actual prednisone use per day was computed as the average over all days in the week.
Time Frame: Baseline to Week 26
Population: Subset of Intent-to-Treat Who Experienced Lesion Cessation
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 5 | 3
mg | 4009.0 (2351.2) | 6446.7 (4225.1)

8. Secondary Outcome: Total Prednisone Dosage Required for Participants to Achieve 80% Healing of Existing Erosions
Description: Each participant's prednisone dose was summed from the time of enrollment until the date of 80% healing of existing erosions. Actual prednisone use per day was computed as the average over all days in the week.
Time Frame: Baseline to Week 26
Population: Subset of Intent-to-Treat Who Experienced Erosion Healing
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 5 | 4
mg | 2921.5 (2978.2) | 2958.8 (3223.4)

9. Secondary Outcome: Participant Health Related Quality of Life (Medical Outcome Study Short Form 36) Score Changes From Baseline to Week 18
Description: The Medical Outcome Study Short Form 36 (MOS SF-36) measures health -related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Change from baseline is computed as the value at Week 18 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value worsening.
Time Frame: Baseline to Week 18
Population: Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 9
units on a scale
  Physical Functioning Scale | 4.0 (12.1) | 4.0 (7.2)
  Role Functioning Scale | 0.3 (14.2) | 6.3 (10.7)
  Bodily Pain Scale | 3.7 (14.8) | 3.2 (12.1)
  General Health Scale | -0.8 (7.1) | 3.6 (5.8)
  Physical Component Scale | 2.2 (8.8) | 3.5 (7.3)
  Vitality Scale | -1.6 (8.1) | 1.7 (10.1)
  Social Functioning Scale | 0.0 (11.5) | 3.0 (13.7)
  Role Emotional Scale | 1.2 (21.5) | 4.8 (13.3)
  Mental Health Scale | 1.4 (6.5) | 6.6 (10.4)
  Mental Component Scale | -0.5 (9.6) | 4.4 (13.3)

10. Secondary Outcome: Participant Dermatology-Related Quality of Life Changes From Baseline to Week 18
Description: The Dermatology Life Quality Index (DLQI) is a 10-question questionnaire with a weighted value to each question. The DLQI score was calculated by summing the score of each question, resulting in a maximum score of 30 and a minimum score of 0. The higher the score, the greater quality of life is impaired. Change from baseline values (defined as the visit value - baseline value) were calculated. A negative change indicates better quality of life; a positive change indicates poorer quality of life.
Time Frame: Baseline to Week 18
Population: Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | -2.0 (3.1) | -4.0 (10.8)

11. Secondary Outcome: Participant Duration of Clinical Response
Description: The primary efficacy endpoint of response to treatment at Week 18 was reassessed at study weeks 22 and 26 for participants who were responders at Week 18. Participants classified as responders had: 1. Achieved a prednisone dosage <= 25% of the initial starting dose or <= 10 mg/day (whichever is greater), and 2. had no new blisters within the previous 4 weeks.
Time Frame: Baseline to Week 26
Population: Participants in the Intent-to-Treat Population Who Were Responders at Week 18
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 1 | 1
Participants
  Week 22 | 1 | 0
  Week 26 | 1 | 0

12. Secondary Outcome: Participants Who Experienced Severe Infusion Reactions
Description: Participants who experienced severe infusion reactions of Grade 3 or greater based on the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0 were assessed.
Time Frame: Baseline to Week 26
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

13. Secondary Outcome: Participants Who Experienced Severe Infectious Complications
Description: Serious and life-threatening infections of Grade 3 or greater based on the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0 were assessed.
Time Frame: Baseline to Week 26
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

14. Secondary Outcome: Adverse Events Resulting in Treatment Discontinuation
Description: Adverse events experienced by participants resulting in study treatment discontinuation and assessed by the investigators as at least possibly related to treatment (i.e., possibly, probably, definitely) were assessed.
Time Frame: Baseline to Week 26
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants | 2 | 2
Statistical Analysis 1: Comparison: Experimental: Infliximab (Remicade, Revellex) vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.3 to 0.3]

15. Secondary Outcome: Participant Pemphigus Vulgaris Disease Activity Score
Description: The Pemphigus Vulgaris Disease Activity (PVDA) score was used to grade a participant's disease activity using the SAGE II computerized burn mapping system, which calculated the total body surface area (BSA) involved. Scores were based on the number of new lesions and blisters present, old lesion history and BSA involved. Scores range from 0 to 3 (none to severe disease activity). A new disease activity score of 3 or an old lesion score of 3 indicates active disease. New disease activity scores of 3 for a 1-month duration or an old lesion score of 3 for 2 consecutive months was cause for removal from the study treatment
Time Frame: Baseline to Week 26
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Experimental: Infliximab (Remicade, Revellex) | Placebo Comparator: Placebo
Number analyzed (Participants) | 10 | 10
Participants
  New Scores of 3 for a 1- Month Duration | 0 | 0
  Old Lesion Scores of 3 in 2 Consecutive Mos. | 0 | 0

ADVERSE EVENTS:
Description: All Adverse Events are included due to low sample size (20 participants).
Groups:
- Infliximab: Subjects randomized to the Infliximab group
- Placebo: Subjects randomized to the Placebo group
Arm/Group | Infliximab | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=10) | Placebo (N=10)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=10) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 3 (3) | 4 (5)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pitting oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (3) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Monocyte count increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (3)
Migraine (Nervous system disorders) | 2 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination, olfactory (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No